CLINICAL TRIAL: NCT04367532
Title: Foam Rolling and Tissue Flossing of the Cuff Muscles: Acute Effect on Jump Height, Sprint Performance and Achilles Tendon Stiffness
Brief Title: Foam Rolling and Tissue Flossing of the Cuff Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Aalborg University (Other); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Sebastian Klich, Dr., Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: USPEWroclaw; 26/2016 (Other: University School of Physical Education in Wroclaw)
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Ankle Injuries; Ankle Sprains
Keywords: self myofascial release; injury prevention; performance; athletic training
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be allocated to intervention (foam rolling, tissue flossing) or control group (without any intervention) using a randomized list of allocated numbers generated by a computer program. Investigator and Outcomes Assessor will be blinded to the allocation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam rolling (Experimental): Foam rolling of cuff muscles.
  Interventions: Other: Foam rolling
- Tissue flossing (Experimental): Tissue flossing of cuff muscles.
  Interventions: Other: Tissue flossing
- Control group (No Intervention): Without any intervention.

INTERVENTIONS:
Other: Foam rolling — Foam rolling performed on cuff muscles in 3 sets of 30 seconds per each muscle part in duration with a 15-second rest between sets. The first sets on the central part of the cuff muscles, the second on the medial and third on the lateral side of the cuff.
  Arms: Foam rolling
Other: Tissue flossing — A standard cuff muscle bandaging technique on cuff muscle. After the application, each participant is asked to perform a 2 min ankle-exercise program.
  Arms: Tissue flossing

SUMMARY:
The hypothesis is that self-myofascial release (SMR) intervention on the cuff muscles would affect positively sprint performance and jump height, as well as, decrease Achilles tendon stiffness. The second hypothesis is that tissue flossing would be more effective than foam rolling.

The participants will be randomly assigned to foam rolling, tissue flossing, and control group (without any intervention). After the intervention, repeated measures will be performed (15m sprint, countermovement jump (CMJ) and Achilles tendon stiffness). This will aim to improve sprint time, jump height and decrease tendon stiffness.

DETAILED DESCRIPTION:
Foam rolling provides beneficial results in ankle range of motion, muscle flexibility or muscle sourness. Tissue flossing is popular in athletic training and physical therapy, as an effective strategy for ankle range of motion or performance. However, there is a lack of knowledge about the use of foam rolling and tissue flossing during a 60 minutes post-intervention examination on the performance and soft tissue stiffness.

The main aim of this study is to investigate the effect of foam rolling and tissue flossing of the cuff on sprint performance, jump height and Achilles tendon stiffness at different time points. The second aim is to assess the effectiveness of those self-myofascial release methods (SMR).

This study will include healthy, recreational active subjects aged between 20 and 25 years old.

ELIGIBILITY:
Inclusion Criteria:

* Regular physical exercise activity (~3 times per week).

Exclusion Criteria:

* Experience with the application of foam rolling and tissue flossing.
* Current or prior pain or injury in the lower extremity.
* Previous history of surgery in the lower extremity.
* Cardiovascular disabilities.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Change in counter-movement jump (CMJ) | Baseline, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes
  A maximum vertical jump with counter-movement.
Change in 15-meter sprint run | Baseline, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes
  The 15-meter sprint involves a participant starting behind a timing gate and running through a second timing gate 15 meters away.
Change in viscoelastic properties of the Achilles tendon. | Baseline, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes
  Stiffness measured on (1) Achilles tendon origin, (2) Achilles tendon on the center ankle joint, and (3) intermuscular septum between medial and lateral head of the gastrocnemius muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kawczyński, Prof., Study Director — University School of Physical Education in Wrocław
Locations (1):
- University Team Sport Hall, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skarabot J, Beardsley C, Stirn I. Comparing the effects of self-myofascial release with static stretching on ankle range-of-motion in adolescent athletes. Int J Sports Phys Ther. 2015 Apr;10(2):203-12. PMID 25883869
- [Background] Smith JC, Pridgeon B, Hall MC. Acute Effect of Foam Rolling and Dynamic Stretching on Flexibility and Jump Height. J Strength Cond Res. 2018 Aug;32(8):2209-2215. doi: 10.1519/JSC.0000000000002321. PMID 29621115
- [Background] Driller M, Mackay K, Mills B, Tavares F. Tissue flossing on ankle range of motion, jump and sprint performance: A follow-up study. Phys Ther Sport. 2017 Nov;28:29-33. doi: 10.1016/j.ptsp.2017.08.081. Epub 2017 Aug 24. PMID 28950149